CLINICAL TRIAL: NCT02218788
Title: An Open-label, Retrospective, Postmarketing Study of Safety and Performance of Hydroxytite, a Calcium Hydroxyapatite Based Filler for Facial Soft Tissue Augmentation.
Brief Title: Injectable Filler for Facial Soft Tissue Augmentation
Status: Completed | Type: Observational
Sponsor: Panaxia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Hydroxytite p100:2013
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Wrinkles
Keywords: Nasolabial folds; Marionette lines; Cheek bones; Jaw lines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the safety and performance of Hydroxytite in all subjects who have received sub dermal or deep dermal injections.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 18 years of age
* Patient received Hydroxytite injection(s).

Exclusion Criteria:

• Patient declines to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients treated with Hydroxytite, above the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety of Hydroxytite (Crystalys) in subjects who received subdermal or deep-dermal injections | 6 months
  Adverse events or Serious adverse events, Injection site reactions.

SECONDARY OUTCOMES:
Performance | 6 months
  To give a score, using the LRS, to Hydroxytite treatment compared to patient's baseline
Performance | 6 months
  To give a score, using the Global Aesthetic Improvement Scale (GAIS), to Hydroxytite treatment compared to patient's baseline